CLINICAL TRIAL: NCT01425996
Title: A Phase I/II, Dose-escalation Study of Lipotecan® Plus Radiotherapy in Locally Advanced Hepatocellular Carcinoma
Brief Title: A Dose-escalation Study of Lipotecan® Plus Radiotherapy in Locally Advanced Hepatocellular Carcinoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Taiwan Liposome Company (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TLC388.2
Record Dates: First submitted 2011-08-15; First posted 2011-08-30 (Estimated); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Carcinoma, Hepatocellular
Keywords: HCC; PVTT
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — TLC 388

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lipotecan® (TLC388) (Experimental): Dosage form: 40mg TLC388 base/vial lyophilized cake Dose: Chemotherapy, i.v. q.w. x 6 doses (dose-escalation)
  * The dosage regimen would be escalated gradually until MTD had been found out.
  Interventions: Drug: Lipotecan® (TLC388)

INTERVENTIONS:
Drug: Lipotecan® (TLC388) — * Cohort A1: TLC388 15 mg/m2 x 6 dose + 3DCRT
  * Cohort A2: TLC388 30 mg/m2 x 6 dose + 3DCRT
  * Cohort A3: TLC388 40 mg/m2 x 6 dose + 3DCRT
  * Cohort A4: TLC388 50 mg/m2 x 6 dose + 3DCRT (dose-escalation)
  * Cohort A"x": TLC388 "MTD" x 6 dose + 3DCRT
  Other Names: Lipotecan (TLC388)

SUMMARY:
Radiotherapy (R/T) for locally advanced hepatocellular carcinoma (HCC) is often used in patient who is not suitable for transarterial chemoembolization (TACE) and other local therapy, especially in those with portal vein tumor thrombosis (PVTT) caused by tumor cells. Several previous studies have showed that local R/T is tolerable and can induce a substantial tumor response in HCC management. In addition, the safety, toxicity and preliminary efficacy of Lipotecan® (TLC388) has also been proved in patients with terminal malignancy. This study aims to evaluate the safety, tolerability and efficacy of concomitant Lipotecan® and radiotherapy in patients with locally advanced HCC and PVTT.

DETAILED DESCRIPTION:
Lipotecan® is a drug product of TLC388 HCl, which is a potent camptothecin analog with cytotoxic activities against a variety of human tumor cell lines and anti-tumor activities in several xenograft models with human tumor cell lines. Structurally, TLC388 HCl is related to other camptothecins, but it has been chemically modified to improve stability and potency, and to minimize toxicities.

ELIGIBILITY:
Inclusion Criteria:

* Females or males 20-70 years of age (inclusive)
* Patients with histological confirmed HCC or other conditions
* Patients with locally advanced HCC and PVTT that is not suitable for other local therapies
* Other inclusion criteria also apply

Exclusion Criteria:

* Females who are pregnant/lactating or planning to be pregnant, or patients of childbearing potential who are not using medically recognized method of contraception.
* Patients with documented extrahepatic metastasis
* Patients with stage III-IV encephalopathy or tense ascites
* Patients who have received any local or systemic therapy for HCC within 4 weeks prior to the initiation of study treatment
* Patients who have received Lipotecan® treatment prior to the initiation of study treatment
* Other exclusion criteria also apply

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2011-10-27 (Actual); Primary Completion 2014-10-03 (Actual); Study Completion 2014-10-03 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | week 12
  Maximum tolerated dose
PVTT response rate | week7
  PVTT response rate
Dose-limiting toxicity (DLT) | week 12
  Dose-limiting toxicity
Adverse Event/Serious Adverse Event | week 12
  Serious/ Adverse Event

SECONDARY OUTCOMES:
Hepatic tumor response rate (overall tumor response rate) | week7, week12
  Hepatic tumor response rate (overall tumor response rate)
Tumor downstaging rate | week7, week12
  Tumor downstaging rate
Time to progression (TTP) | week7, week12, 1 year
  Time to progression
Progression-free survival (PFS) | week7, week12, 1 year
  Progression-free survial
Overall survival (OS) | week7, week12, 1year
  Overall survival
Change from baseline in tumor marker/biomarkers | week4, week7, week12
  Change from baseline in tumor marker/biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: Tsang-En Wa, MD, Principal Investigator — Mackay Memorial Hospital; Yee Chao, MD, Principal Investigator — Taipei Veteran General Hospital; Chen-Hsi Hsieh, MD, Principal Investigator — Far Eastern Memorial Hospital; Jacqueline Whang-Peng, MD, Principal Investigator — Wan Fang Hospital
Locations (2):
- Taiwan (2):
  - Mackay Memorial Hospital, Taipei
  - Taipei Veteran General Hospital, Taipei